CLINICAL TRIAL: NCT02577354
Title: ReActiv8 Implantable Neurostimulation System for Chronic Low Back Pain (ReActiv8-B)
Brief Title: ReActiv8 Implantable Neurostimulation System for Chronic Low Back Pain
Acronym: ReActiv8-B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mainstay Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 950057
Record Dates: First submitted 2015-10-12; First posted 2015-10-16 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental)
  Interventions: Device: ReActiv8 Implantable Stimulation System (Patient Appropriate Stimulation)
- Control (Experimental)
  Interventions: Device: ReActiv8 Implantable Stimulation System (Low Stimulation)

INTERVENTIONS:
Device: ReActiv8 Implantable Stimulation System (Patient Appropriate Stimulation) — ReActiv8 implanted and configured to deliver stimulation at a patient-appropriate level, and participants instructed to deliver stimulation in two 30-minute sessions per day.
  Arms: Treatment
Device: ReActiv8 Implantable Stimulation System (Low Stimulation) — ReActiv8 implanted and configured to deliver low stimulation, and participants instructed to deliver stimulation in two 30-minute sessions per day.
  Arms: Control

SUMMARY:
The purpose of this trial is to evaluate the safety and efficacy of ReActiv8 for the treatment of adults with Chronic Low Back Pain when used in conjunction with medical management.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥22 years, ≤75 years
2. Chronic Low Back Pain that has persisted >90 days prior to the baseline visit.
3. Continuing low back pain despite >90 days of medical management.
4. Qualifying pain score.
5. Qualifying disability score.
6. Evidence of lumbar multifidus muscle dysfunction.
7. Be willing and capable of giving Informed Consent.
8. Ability to comply with the instructions for use and to operate ReActiv8, and to comply with this Clinical Investigation Plan.
9. Suitable for ReActiv8 surgery as determined by the implanting physician prior to inclusion.

Exclusion Criteria:

1. BMI > 35
2. Back Pain characteristics:

   1. Any surgical correction procedure for scoliosis at any time, or a current clinical diagnosis of scoliosis.
   2. Lumbar spine stenosis, as defined by an anterior-posterior diameter of the spinal canal of <10mm in subjects with lower extremity pain.
   3. Neurological deficit possibly associated with the back pain (e.g. foot drop).
   4. Back pain due to pelvic or visceral reasons (e.g.: endometriosis or fibroids) or infection (e.g.: post herpetic neuralgia).
   5. Back pain due to inflammation or damage to the spinal cord or adjacent structures (e.g. arachnoiditis or syringomyelia).
   6. Pathology seen on MRI that is clearly identified and is likely the cause of the CLBP that is amenable to surgery.
   7. Back pain due to vascular causes such as aortic aneurysm and dissection.
3. Any current indication for back surgery according to local institutional guidelines, or has indication for back surgery but cannot undergo surgery for other reasons.
4. Leg pain described as being worse than back pain, or radiculopathy (neuropathic pain) below the knee.
5. Source of pain is the sacroiliac joint as determined by the Investigator.
6. Drug use.
7. Surgical and other procedures exclusions.
8. Any prior diagnosis of lumbar vertebral compression fracture, lumbar pars fracture, or lumbar annular tear with disc protrusion that is amenable to surgery.
9. Planned surgery.
10. Co-morbid chronic pain conditions.
11. Other clinical conditions.
12. Psycho-social exclusions.
13. Protocol compliance exclusions.
14. General exclusions.

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2016-08; Primary Completion 2018-11 (Actual); Study Completion 2024-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Gilligan, MD, MBA, Study Chair — Brigham and Women's Hospital
Locations (26):
- United States (16):
  - University of California, San Diego, La Jolla, California
  - The Spine Institute, Santa Monica, California
  - University of Colorado Hospital, Aurora, Colorado
  - Indiana Spine Group, Carmel, Indiana
  - OrthoIndy, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - The Brigham and Women's Hospital, Boston, Massachusetts
  - Beaumont Health, Royal Oak, Michigan
  - Duke University Medical Center, Durham, North Carolina
  - Center for Clinical Research, Winston-Salem, North Carolina
  - Louis Stokes VA Medical Center, Cleveland, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - Upstate Clinical Trials, Spartanburg, South Carolina
  - Northwest Orthopaedic Specialists, Spokane, Washington
  - Center for Pain Relief, Charleston, West Virginia
- Australia (4):
  - Genesis Research Services, Broadmeadow, New South Wales
  - Sunshine Coast Clinical Research, Noosa, Queensland
  - Pain Medicine of South Australia, Welland, South Australia
  - Monash Clinical Research, Clayton, Victoria
- Belgium (2):
  - AZ Nikolaas, Sint-Niklaas
  - Sint Augustinus, Wilrijk
- Erasmus MC University Medical Center, Rotterdam, Netherlands
- United Kingdom (3):
  - Seacroft Hospital, Leeds
  - St. Bartholomew's Hospital, London
  - The James Cook University Hospital, Middlesbrough

REFERENCES:
- [Background] Gilligan C, Burnside D, Grant L, Yong RJ, Mullins PM, Schwab F, Mekhail N. ReActiv8 Stimulation Therapy vs. Optimal Medical Management: A Randomized Controlled Trial for the Treatment of Intractable Mechanical Chronic Low Back Pain (RESTORE Trial Protocol). Pain Ther. 2023 Apr;12(2):607-620. doi: 10.1007/s40122-023-00475-4. Epub 2023 Feb 14. PMID 36787013
- [Result] Gilligan C, Volschenk W, Russo M, Green M, Gilmore C, Mehta V, Deckers K, De Smedt K, Latif U, Georgius P, Gentile J, Mitchell B, Langhorst M, Huygen F, Baranidharan G, Patel V, Mironer E, Ross E, Carayannopoulos A, Hayek S, Gulve A, Van Buyten JP, Tohmeh A, Fischgrund J, Lad S, Ahadian F, Deer T, Klemme W, Rauck R, Rathmell J, Levy R, Heemels JP, Eldabe S; ReActiv8-B investigators. An implantable restorative-neurostimulator for refractory mechanical chronic low back pain: a randomized sham-controlled clinical trial. Pain. 2021 Oct 1;162(10):2486-2498. doi: 10.1097/j.pain.0000000000002258. PMID 34534176
- [Result] Gilligan C, Volschenk W, Russo M, Green M, Gilmore C, Mehta V, Deckers K, De Smedt K, Latif U, Georgius P, Gentile J, Mitchell B, Langhorst M, Huygen F, Baranidharan G, Patel V, Mironer E, Ross E, Carayannopoulos A, Hayek S, Gulve A, Van Buyten JP, Tohmeh A, Fischgrund J, Lad S, Ahadian F, Deer T, Klemme W, Rauck R, Rathmell J, Maislin G, Heemels JP, Eldabe S; ReActiv8-B Investigators. Long-Term Outcomes of Restorative Neurostimulation in Patients With Refractory Chronic Low Back Pain Secondary to Multifidus Dysfunction: Two-Year Results of the ReActiv8-B Pivotal Trial. Neuromodulation. 2023 Jan;26(1):87-97. doi: 10.1016/j.neurom.2021.10.011. Epub 2021 Dec 18. PMID 35088722
- [Result] Gilligan C, Volschenk W, Russo M, Green M, Gilmore C, Mehta V, Deckers K, De Smedt K, Latif U, Sayed D, Georgius P, Gentile J, Mitchell B, Langhorst M, Huygen F, Baranidharan G, Patel V, Mironer E, Ross E, Carayannopoulos A, Hayek S, Gulve A, Van Buyten JP, Tohmeh A, Fischgrund J, Lad S, Ahadian F, Deer T, Klemme W, Rauck R, Rathmell J, Schwab F, Maislin G, Heemels JP, Eldabe S. Three-Year Durability of Restorative Neurostimulation Effectiveness in Patients With Chronic Low Back Pain and Multifidus Muscle Dysfunction. Neuromodulation. 2023 Jan;26(1):98-108. doi: 10.1016/j.neurom.2022.08.457. Epub 2022 Sep 27. PMID 36175320
- [Result] Gilligan C, Volschenk W, Russo M, Green M, Gilmore C, Mehta V, Deckers K, De Smedt K, Latif U, Sayed D, Georgius P, Gentile J, Mitchell B, Langhorst M, Huygen F, Baranidharan G, Patel V, Mironer E, Ross E, Carayannopoulos A, Hayek S, Gulve A, Van Buyten JP, Tohmeh A, Fischgrund J, Lad S, Ahadian F, Deer T, Klemme W, Rauck R, Rathmell J, Maislin G, Heemels JP, Eldabe S. Five-Year Longitudinal Follow-Up of Restorative Neurostimulation Shows Durability of Effectiveness in Patients With Refractory Chronic Low Back Pain Associated With Multifidus Muscle Dysfunction. Neuromodulation. 2024 Jul;27(5):930-943. doi: 10.1016/j.neurom.2024.01.006. Epub 2024 Mar 12. PMID 38483366
- [Derived] Shaffrey C, Gilligan C. Effect of Restorative Neurostimulation on Major Drivers of Chronic Low Back Pain Economic Impact. Neurosurgery. 2023 Apr 1;92(4):716-724. doi: 10.1227/neu.0000000000002305. Epub 2023 Feb 14. PMID 36786565

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: ReActiv8 Implantable Stimulation System (patient appropriate stimulation): ReActiv8 implanted and configured to deliver stimulation at a patient-appropriate level and participants instructed to deliver stimulation in two 30-minute sessions per day.
- Control/Crossover: ReActiv8 Implantable Stimulation System (low stimulation): ReActiv8 implanted and configured to deliver low stimulation, and participants instructed to deliver stimulation in two 30-minute sessions per day.
  After 120 day visit, participants crossed over to have their device programmed to deliver stimulation at a patient-appropriate level.
Period: Overall Study
Arm/Group | Treatment | Control/Crossover
Started | 102 | 102
120 Day Primary Endpoint (Three participants in total lost to follow-up) | 100 | 101
Completed (Completed 1 year follow-up for FDA PMA report (a minimum of 150 participants required)) | 87 | 89
Not Completed | 15 | 13
Not completed — Lack of Efficacy | 4 | 4
Not completed — Lost to Follow-up | 3 | 1
Not completed — Missed Visit | 4 | 3
Not completed — Adverse Event | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Control/Crossover: ReActiv8 Implantable Stimulation System (low stimulation): ReActiv8 implanted and configured to deliver low stimulation, and participants instructed to deliver stimulation in two 30-minute sessions per day.
  After the 120-day visit, participants crossed over to have their device programmed to deliver stimulation at a patient-appropriate level.
- Total: Total of all reporting groups
Arm/Group | Treatment | Control/Crossover | Total
Number analyzed (Participants) | 102 | 102 | 204
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (10) | 48 (9) | 47 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 54 | 110
  Male | 46 | 48 | 94
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 97 | 95 | 192
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 96 | 96 | 192
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  Netherlands | 2 | 4 | 6
  Belgium | 9 | 8 | 17
  United States | 42 | 43 | 85
  United Kingdom | 13 | 12 | 25
  Australia | 36 | 35 | 71
BMI [Mean (Standard Deviation); unit: Kg/m^2] | 28 (4) | 28 (4) | 28 (4)
Pain Duration (years from onset) [Mean (Standard Deviation); unit: years] | 14.4 (10.8) | 13.9 (10.4) | 14.2 (10.6)
Percent of Days with Low Back Pain [Mean (Standard Deviation); unit: percent] — Participant report of percent of days in the past 12 months with low back pain.
  percent | 97 (8) | 97 (8) | 97 (8)
Evidence of Leg Pain [Count of Participants; unit: Participants] — Participant report of current leg pain.
  Participants | 32 | 30 | 62
Number of Prior Physical Therapy Sessions [Mean (Standard Deviation); unit: sessions] | 30 (39) | 32 (63) | 31 (52)
Previous Rhizotomy [Count of Participants; unit: Participants] | 8 | 17 | 25
Previous Injection Procedures [Count of Participants; unit: Participants] — Injection procedures refers to epidural procedures (e.g., spinal block)
  Participants | 53 | 46 | 99
VAS for Low Back Pain [Mean (Standard Deviation); unit: units on a scale] — The instrument used for evaluating pain is the continuous Visual Analog Scale (VAS) comprised of a horizontal line 10 cm in length, anchored by 2 verbal descriptors, where zero indicates no pain and 10 indicates worst imaginable pain. The value reported is a 7-day average low back pain.
  units on a scale | 7.3 (.7) | 7.2 (.7) | 7.3 (.7)
Oswestry Disability Index [Mean (Standard Deviation); unit: units on a scale] — ODI is reported as a score from 0 to 100%, where 0%-20% indicates minimal disability, 21%-40% indicates moderate disability, 41%-60% indicates severe disability, 61%-80% indicates crippled, and 81%-100% indicates bedbound or an exaggeration of symptoms.
  units on a scale | 40 (10) | 38 (10) | 39 (10)
EQ-5D-5L Index Score [Mean (Standard Deviation); unit: units on a scale] — The EQ-5D Index is scored on a scale of -0.594 to 1.00, with a score of 1.00 indicating full health.
  units on a scale | 0.572 (0.182) | 0.598 (0.165) | 0.585 (0.174)
Low Back Pain Medications of Any Type [Count of Participants; unit: Participants] | 77 | 85 | 162
Opioid Use [Count of Participants; unit: Participants] | 36 | 40 | 76

OUTCOME MEASURES:

1. Primary Outcome: Responder Rate of Low Back Pain With No Increase in Pain Medications
Description: Comparison of responder rates for low back pain VAS between Treatment and Control groups.
  The Primary Efficacy Endpoint is a comparison of responder rates between Treatment and Control groups, where a "responder" is a participant with ≥30% reduction from baseline in average low back pain VAS, without any increase from baseline in pain medications and/or muscle relaxants for any reason including non low back pain reasons.
  The instrument used for evaluating pain is the continuous Visual Analog Scale (VAS) comprised of a horizontal line 10 cm in length, anchored by 2 verbal descriptors, where zero indicates no pain and 10 indicates worst imaginable pain. The value reported is a 7-day average low back pain.
  Any increase in dosage of a pain medication or any new pain medication taken for any reason counts as an increase in medications.
Time Frame: 120 Days
Population: 100 treatment group participants and 101 control group participants returned for the 120 day visit. Results for the 3 participants lost to follow-up were included using multiple imputation.
Measure: Number; unit: percentage of responsers
Groups:
- Treatment: ReActiv8 Implantable Stimulation System (patient-appropriate stimulation): ReActiv8 implanted and configured to deliver stimulation at a patient-appropriate level, and participants instructed to deliver stimulation in two 30-minute sessions per day.
Arm/Group | Treatment | Control
Number analyzed (Participants) | 102 | 102
percentage of responsers | 57.1 | 46.6
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority; p = 0.138, Wald asymptotic test of proportions — The threshold for statistical significance was p=0.05; Cui p-value adjustment for sample size re-estimation at interim analysis; Multiple imputation utilized for 3 participants lost to follow-up

2. Primary Outcome: Mean Change in Low Back Pain VAS
Description: Comparison of change in LBP VAS (120 days from baseline) between the Treatment and Control groups. The instrument used for evaluating pain is the continuous Visual Analog Scale (VAS) comprised of a horizontal line 10 cm in length, anchored by 2 verbal descriptors, where zero indicates no pain and 10 indicates worst imaginable pain. The value reported is a 7-day average low back pain.
  A change to a lower score (negative value) indicates improvement.
Time Frame: 120 Days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 100 | 101
score on a scale | -3.3 (2.7) | -2.4 (2.9)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority; p = 0.032, t-test, 2 sided — Threshold for statistical significance was p=0.05

3. Primary Outcome: Cumulative Proportion of Responders Analysis (CPRA) for the Primary Endpoint to Compare Participants Responses Over a Full Range of Response Levels
Description: The CPRA, which was prespecified in the clinical protocol and statistical analysis plan prior to the start of the trial, was performed using the same data as used for the primary endpoint analysis and was included as part of the primary endpoint analysis
Time Frame: 120 Days
Population: 3 participants lost to follow-up included using multiple imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 102 | 102
percentage of participants
  >0% Reduction in Pain | 83.0 | 71.3
  >10% Reduction in Pain | 78.0 | 63.4
  >20% Reduction in Pain | 68.0 | 50.5
  >30% Reduction in Pain | 57.0 | 46.5
  >40% Reduction in Pain | 51.0 | 39.6
  >50% Reduction in Pain | 42.0 | 33.7
  >60% Reduction in Pain | 36.0 | 30.7
  >70% Reduction in Pain | 28.0 | 24.8
  >80% Reduction in Pain | 24.0 | 19.8
  >90% Reduction in Pain | 16.0 | 11.9
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority; p = 0.0499, Friedman's regression analysis — The threshold for significance was p=0.05; Multiple Imputation utilized for 3 participants lost to follow-up

4. Primary Outcome: Serious Device and/or Procedure Related Adverse Event Rate
Description: The primary safety assessment is of serious device and/or procedure related adverse events in all participants at 120 days.
  The 8 events reported below are 6 implant site pocket infections, 1 intra-operative upper airway obstruction, and 1 non-radicular, focal numbness on the surface of the thigh.
Time Frame: 120 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 102 | 102
Participants | 3 | 5

5. Secondary Outcome: Change in Oswestry Disability Index (ODI)
Description: Comparison of change in ODI (120 days from baseline) between Treatment and Control groups. ODI is reported as a score from 0 to 100%, where 0%-20% indicates minimal disability, 21%-40% indicates moderate disability, 41%-60% indicates severe disability, 61%-80% indicates crippled, and 81%-100% indicates bedbound or an exaggeration of symptoms.
  A change to a lower score (negative value) indicates improvement.
Time Frame: 120 Days
Population: Completers Analysis. Three participants (2 Treatment, 1 Control) were lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 100 | 101
score on a scale | -17.5 (15.1) | -12.2 (14.6)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority; p = 0.011, t-test, 2 sided — Threshold for statistical significance was p=0.05

6. Secondary Outcome: Change in European Quality of Life Score on Five Dimensions (EQ-5D)
Description: Comparison of change in EQ-5D (120 days from baseline) between Treatment and Control groups. The EQ-5D Index is scored on a scale of -0.594 to 1.00, with a score of 1.00 indicating full health.
  A change to a higher score (positive value) indicates improvement.
Time Frame: 120 Days
Population: Completers Analysis. Three participants (2 Treatment, 1 Control) were lost to follow-up. An additional patient in the Control group did not complete the questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 100 | 100
score on a scale | 0.186 (0.199) | 0.115 (0.178)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority; p = 0.009, t-test, 2 sided — Threshold for statistical significance was p=0.05

7. Secondary Outcome: Change in Percent Pain Relief (PPR)
Description: PPR is a patient-reported percent of pain relief at 120 days compared to the pain at baseline, where 0% indicates no pain relief compared to baseline, and 100% indicates complete pain relief compared to baseline.
Time Frame: 120 Days
Population: Completers Analysis. Three participants (2 Treatment, 1 Control) were lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 100 | 101
score on a scale | 52 (32) | 35 (36)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority; p < 0.001, t-test, 2 sided — Threshold for statistical significance was 0.05

8. Secondary Outcome: Subject Global Impression of Change (SGIC)
Description: A questionnaire completed with the following item: Since I enrolled in the study, my overall status is 1) Very much improved, 2) Much improved, 3) Minimally improved, 4) No change, 5) Minimally worse, 6) Much worse, 7) Very much worse
Time Frame: 120 Days
Population: Completers Analysis. Three participants (2 Treatment, 1 Control) were lost to follow-up.
Measure: Number; unit: participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 100 | 101
participants
  Much Better | 32 | 18
  Better | 22 | 16
  A Little Better | 25 | 29
  No Change | 10 | 24
  A Little Worse | 6 | 5
  Worse | 4 | 6
  Much Worse | 1 | 3
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority; p = 0.003, Wilcoxon (Mann-Whitney) — Threshold for statistical significance was p=0.05

9. Secondary Outcome: Resolution of Back Pain (VAS ≤2.5 cm)
Description: Resolution of back pain (remitter rate) was defined as a participant with 7-day average low back pain VAS ≤2.5 cm on the 10 cm VAS.
Time Frame: 120 Days
Population: Completers Analysis. Three participants (2 Treatment, 1 Control) were lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 100 | 101
Participants | 34 | 28
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority; p = 0.335, Chi-squared — Threshold for statistical significance was p=0.05

10. Secondary Outcome: LBP VAS Responder Rate at One Year
Description: A "responder" is a participant with ≥30% reduction from baseline in average low back pain VAS, without any increase from baseline in pain medications and/or muscle relaxants for any reason including non low back pain reasons.
  After the 120 day visit, participants crossed over to have their device programmed to deliver stimulation at a patient-appropriate level. At the one-year time point, participants in the Control/Crossover group have received 8 months of patient-appropriate therapy.
Time Frame: 1 Year
Population: Participants with data at one year.
Measure: Count of Participants; unit: Participants
Groups:
- All (Treatment and Control/Crossover Combined): At the 1-year visit, all participants are receiving patient-appropriate therapy (1 year of patient-appropriated therapy for the Treatment Group, and 8 months of patient-appropriate therapy for the Control Group). This column provides the results for all participants in one group.
Arm/Group | Treatment | Control/Crossover | All (Treatment and Control/Crossover Combined)
Number analyzed (Participants) | 87 | 89 | 176
Participants | 58 | 57 | 115

11. Secondary Outcome: Mean Change in LBP VAS at One Year
Description: Change in LBP VAS at 1 year compared to baseline. The instrument used for evaluating pain is the continuous Visual Analog Scale (VAS) comprised of a horizontal line 10 cm in length, anchored by 2 verbal descriptors, one for each symptom extreme for Low Back Pain. Zero indicates no pain and 10 indicates worst imaginable pain. The value reported is a 7-day average low back pain.
  After the 120 day visit, participants crossed over to have their device programmed to deliver stimulation at a patient-appropriate level. At the one-year time point, participants in the Control/Crossover group have received 8 months of patient-appropriate therapy.
  A change to a lower score (negative value) indicates improvement.
Time Frame: 1 Year
Population: Participants with data at one year.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- All (Treatment and Control/Crossover Combined): At the 1-year visit, all participants are receiving patient-appropriate therapy (1 year of patient-appropriated therapy for the Treatment Group, and 8 months of patient-appropriate therapy for the Control/Crossover Group). This column provides the results for all participants in one group.
Arm/Group | Treatment | Control/Crossover | All (Treatment and Control/Crossover Combined)
Number analyzed (Participants) | 87 | 89 | 176
score on a scale | -4.2 (2.7) | -4.3 (2.5) | -4.3 (2.6)

12. Secondary Outcome: Change in Oswestry Disability Index (ODI) at One Year
Description: Change in ODI at 1 year compared to baseline. ODI is reported as a score from 0 to 100%, where 0%-20% indicates minimal disability, 21%-40% indicates moderate disability, 41%-60% indicates severe disability, 61%-80% indicates crippled, and 81%-100% indicates bedbound or an exaggeration of symptoms.
  After the 120 day visit, participants crossed over to have their device programmed to deliver stimulation at a patient-appropriate level. At the one-year time point, participants in the Control/Crossover group have received 8 months of patient-appropriate therapy.
  A change to a lower score (negative value) indicates improvement.
Time Frame: 1 Year
Population: Participants with data at one year.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control/Crossover | All (Treatment and Control/Crossover Combined)
Number analyzed (Participants) | 87 | 89 | 176
score on a scale | -20.1 (17.2) | -19.8 (14.5) | -19.9 (15.8)

13. Secondary Outcome: Change in European Quality of Life Score on Five Dimensions (EQ-5D) at One Year
Description: Change in EQ-5D at 1 year compared to baseline. The EQ-5D Index is scored on a scale of -0.594 to 1.00, with a score of 1.00 indicating full health.
  After the 120 day visit, participants crossed over to have their device programmed to deliver stimulation at a patient-appropriate level. At the one-year time point, participants in the Control/Crossover group have received 8 months of patient-appropriate therapy.
  A change to a higher score (positive value) indicates improvement.
Time Frame: 1 Year
Population: Participants with data at one year.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control/Crossover | All (Treatment and Control/Crossover Combined)
Number analyzed (Participants) | 87 | 89 | 176
score on a scale | 0.210 (0.235) | 0.187 (0.177) | 0.198 (0.207)

14. Secondary Outcome: Percent Pain Relief at One Year
Description: PPR is a patient-reported percent of pain relief compared to the pain at baseline, where 0% indicates no pain relief compared to baseline, and 100% indicates complete pain relief compared to baseline.
  After the 120 day visit, participants crossed over to have their device programmed to deliver stimulation at a patient-appropriate level. At the one-year time point, participants in the Control/Crossover group have received 8 months of patient-appropriate therapy.
Time Frame: 1 Year
Population: Participants with data at one year.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control/Crossover | All (Treatment and Control/Crossover Combined)
Number analyzed (Participants) | 87 | 89 | 176
score on a scale | 65 (33) | 66 (33) | 66 (32)

15. Secondary Outcome: Subject Global Impression of Change (SGIC) at One Year
Description: A questionnaire with the following item: Since I enrolled in the study, my overall status is 1) Very much improved, 2) Much improved, 3) Minimally improved, 4) No change, 5) Minimally worse, 6) Much worse, 7) Very much worse
  After the 120 day visit, participants crossed over to have their device programmed to deliver stimulation at a patient-appropriate level. At the one-year time point, participants in the Control/Crossover group have received 8 months of patient-appropriate therapy.
Time Frame: 1 Year
Population: Participants with data at one year.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control/Crossover | All (Treatment and Control/Crossover Combined)
Number analyzed (Participants) | 87 | 89 | 176
Participants
  Much Better | 44 | 40 | 84
  Better | 19 | 23 | 42
  A Little Better | 14 | 14 | 28
  No Change | 6 | 8 | 14
  A Little Worse | 2 | 2 | 4
  Worse | 1 | 1 | 2
  Much Worse | 1 | 1 | 2

16. Secondary Outcome: Resolution of Back Pain at One Year
Description: Resolution of back pain (remitter rate) was defined as a participant with 7-day average low back pain VAS ≤2.5 cm on the 10 cm VAS.
  After the 120 day visit, participants crossed over to have their device programmed to deliver stimulation at a patient-appropriate level. At the one-year time point, participants in the Control/Crossover group have received 8 months of patient-appropriate therapy.
Time Frame: 1 Year
Population: Participants with data at one year.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control/Crossover | All (Treatment and Control/Crossover Combined)
Number analyzed (Participants) | 87 | 89 | 176
Participants | 42 | 49 | 91

17. Other Pre Specified Outcome: Supplementary Analysis of Primary Endpoint: Responder Rate of Low Back Pain With No Increase in Low Back Pain Medications
Description: This pre-specified analysis of the primary endpoint examines the impact of rescue medications taken for acute pain conditions for reasons other than low back pain, by excluding those participants from the analysis who took rescue medications for reasons other than low back pain.
  Nine participants in both groups increased pain medications. In the control group, all nine participants increased pain medications due to low back pain. In the treatment group, three of the nine participants increased pain medications due to low back pain, while six of the nine participants increased pain medications for reasons other than low back pain. Since any increase in pain medications automatically considers a participant a non-responder, these six participants are removed from this analysis to eliminate the confounding factor of increases in pain medications for reasons other than low back pain.
Time Frame: 120 Days
Population: Responder rate (≥30% reduction in low back pain VAS and no increase in pain medications). Six participants with increases in pain medications for reasons other than low back pain are removed from this analysis.
Measure: Number; unit: percentage of responders
Arm/Group | Treatment | Control
Number analyzed (Participants) | 96 | 102
percentage of responders | 60.6 | 46.7
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority; p = 0.048, Wald asymptotic test of proportions — The threshold for statistical significance was p=0.05; Multiple imputation used for three participants lost to follow-up

18. Other Pre Specified Outcome: Treatment Satisfaction
Description: The Treatment Satisfaction Questionnaire asking the participant if they are satisfied with the treatment.
Time Frame: 120 Days
Population: Completers Analysis. Three participants (2 Treatment, 1 Control) were lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 100 | 101
Participants
  Definitely Yes | 61 | 40
  Maybe | 29 | 37
  Definitely Not | 10 | 24
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-value for "Satisfied with Treatment". Threshold for statistical significance was p=0.05

19. Other Pre Specified Outcome: Treatment Satisfaction at One Year
Description: The Treatment Satisfaction Questionnaire asking the participant if they are satisfied with the outcome of the treatment.
  After the 120 day visit, participants crossed over to have their device programmed to deliver stimulation at a patient-appropriate level. At the one-year time point, participants in the Control/Crossover group have received 8 months of patient-appropriate therapy.
Time Frame: 1 Year
Population: Participants with data at one year.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control/Crossover | All (Treatment and Control/Crossover Combined)
Number analyzed (Participants) | 86 | 88 | 174
Participants
  Definitely Yes | 68 | 68 | 136
  Maybe | 12 | 17 | 29
  Definitely Not | 6 | 3 | 9

20. Other Pre Specified Outcome: Clinical Global Impression of Change
Description: Clinical Global Impression consists of the following question completed by the Investigator prior to unblinding: In your opinion as a clinician, compared to the patient's situation at baseline, would you say the patient is: 1) Much better, 2) Slightly better, 3) About the same, 4) Slightly worse, 5) Much worse.
Time Frame: 120 Days
Population: Completers Analysis. Three participants were lost to follow-up (2 Treatment, 1 Control). The questionnaire was not completed for an additional participant in the Control group.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 100 | 100
Participants
  Much Better | 57 | 22
  Slightly Better | 26 | 29
  About the Same | 16 | 42
  Slightly Worse | 1 | 5
  Much Worse | 0 | 2
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Threshold for statistical significance was p=0.05

21. Other Pre Specified Outcome: Clinical Global Impression of Change at One Year
Description: Clinical Global Impression consists of the following question completed by the Investigator prior to unblinding: In your opinion as a clinician, compared to the patient's situation at baseline, would you say the patient is: 1) Much better, 2) Slightly better, 3) About the same, 4) Slightly worse, 5) Much worse.
  After the 120 day visit, participants crossed over to have their device programmed to deliver stimulation at a patient-appropriate level. At the one-year time point, participants in the Control/Crossover group have received 8 months of patient-appropriate therapy.
Time Frame: 1 Year
Population: Participants with data at one year.
Measure: Count of Participants; unit: Participants
Groups:
- All (Treatment and Control/Crossover Combined): At the 1 Year visit, all participants are receiving patient-appropriate therapy (1 year of patient-appropriated therapy for the Treatment Group, and 8 months of patient-appropriate therapy for the Control/Crossover Group). This column provides the results for all participants in one group.
Arm/Group | Treatment | Control/Crossover | All (Treatment and Control/Crossover Combined)
Number analyzed (Participants) | 87 | 89 | 176
Participants
  Much Better | 66 | 63 | 129
  Slightly Better | 11 | 15 | 26
  About the Same | 8 | 10 | 18
  Slightly Worse | 1 | 1 | 2
  Much Worse | 1 | 0 | 1

22. Other Pre Specified Outcome: Change in Opioid Use for Treatment of Low Back Pain at One-Year
Description: Any increase or decrease of dosage or frequency of an opioid taken for the treatment of low back pain was considered a change.
Time Frame: 1 Year
Population: Participants with data at one year who were on opioids at baseline. Since changes in opioids are evaluated only at 1 year (and not compared between groups at 120 days), and all participants are receiving therapy at the 1 year time point, there is no between group comparison. Therefore, the groups are combined for this analysis.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants Combined: At the 1-year visit, all participants are receiving patient-appropriate therapy (1 year of patient-appropriate therapy for the Treatment Group, and 8 months of patient-appropriate therapy for the Control Group).
Arm/Group | All Participants Combined
Number analyzed (Participants) | 65
Participants
  Discontinued or Decreased | 31
  No Change | 29
  Increased or Added | 5

ADVERSE EVENTS:
Time Frame: Events were collected through the 120 day primary endpoint and through one year per the Investigational Device Exemption (IDE). The FDA required a minimum of 150 participants through one year prior to Premarket Approval (PMA) application. These results are adverse events (related and unrelated) reported through the one year visit.
Description: All adverse events were adjudicated by a Clinical Events Committee comprised of independent physicians. The committee adjudicated the type of event, severity of event, and relatedness to the system or procedure.
Groups:
- Treatment -- Blinded Phase (0-120 Days); Treatment -- Open Label Phase (121-365 Days): ReActiv8 Implantable Stimulation System (patient appropriate stimulation): ReActiv8 implanted and configured to deliver stimulation at a patient-appropriate level and participants instructed to deliver stimulation in two 30-minute sessions per day.
- Control -- Blinded Phase (0-120 Days); Crossover -- Open Label Phase (121-365 Days): ReActiv8 Implantable Stimulation System (low stimulation): ReActiv8 implanted and configured to deliver low stimulation, and participants instructed to deliver stimulation in two 30-minute sessions per day.
  After 120 day visit, participants crossed over to have their device programmed to deliver stimulation at a patient-appropriate level.
Arm/Group | Treatment -- Blinded Phase (0-120 Days) | Control -- Blinded Phase (0-120 Days) | Treatment -- Open Label Phase (121-365 Days) | Crossover -- Open Label Phase (121-365 Days)
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/102 | 0/99 | 0/99
Serious Adverse Events (participants affected / at risk) | 4/102 | 6/102 | 3/99 | 2/99
Other Adverse Events (participants affected / at risk) | 32/102 | 24/102 | 25/99 | 34/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment -- Blinded Phase (0-120 Days) (N=102) | Control -- Blinded Phase (0-120 Days) (N=102) | Treatment -- Open Label Phase (121-365 Days) (N=99) | Crossover -- Open Label Phase (121-365 Days) (N=99)
Implant site pocket infection (Injury, poisoning and procedural complications) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Intra-operative airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Numbness in Leg (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute appendicitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Ankle Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest Pain (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Concussion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gallstones (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant Melanoma stage IV (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment -- Blinded Phase (0-120 Days) (N=102) | Control -- Blinded Phase (0-120 Days) (N=102) | Treatment -- Open Label Phase (121-365 Days) (N=99) | Crossover -- Open Label Phase (121-365 Days) (N=99)
Implant site pocket pain/discomfort (Injury, poisoning and procedural complications) | 11 (12) | 11 (11) | 3 (3) | 10 (11)
Device overstimulation of tissue (Product Issues) | 7 (7) | 0 (0) | 5 (6) | 12 (13) — Discomfort associated with stimulation, often related to the titration of therapy and typically resolved with reprogramming.
Back Pain Aggravated (Musculoskeletal and connective tissue disorders) | 11 (11) | 13 (14) | 13 (13) | 17 (17)
Upper Respiratory Infection (Infections and infestations) | 9 (9) | 5 (5) | 5 (5) | 1 (1)
Pain in Hip (Musculoskeletal and connective tissue disorders) | 7 (7) | 0 (0) | 3 (3) | 2 (2)

LIMITATIONS AND CAVEATS:
Dichotomization of primary endpoint reduced statistical power by losing information on exact response magnitude. This limitation is addressed by the cumulative proportion of responders analysis of the primary endpoint data (Outcome Measure #3).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-03-25): https://cdn.clinicaltrials.gov/large-docs/54/NCT02577354/Prot_000.pdf
  • Statistical Analysis Plan (2015-12-10): https://cdn.clinicaltrials.gov/large-docs/54/NCT02577354/SAP_001.pdf